CLINICAL TRIAL: NCT01216371
Title: Prospektiv Randomisierte Multizentrische Phase II-Studie Zur Metastasenresektion Von Lungenfiliae (Poor-prognosis) Beim Klarzelligen Nierenzellkarzinom +/- Adjuvante Sunitinibtherapie über 1 Jahr SMAT - AN 20/04 Der AUO
Brief Title: Resection of Pulmonary Metastasis in Clear Cell Renal Cell Carcinoma +/-Adjuvant Sunitinib Therapy (SMAT)
Acronym: SMAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association of Urologic Oncology (AUO) (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Heidrun Rexer, Priv. Doz. Dr. med. Susanne Krege, urological hospital of Maria Hilf Krankenhaus Krefeld, Association of Urologic Oncology (AUO)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN 20/04; 2008-007609-36 (EudraCT Number)
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Renal Cell Carcinoma; Pulmonary Metastases
Keywords: carcinoma; metastases; renal; lung
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib (Active Comparator): one year adjuvant treatment with sunitinib
  Interventions: Drug: Sunitinib
- Placebo (Placebo Comparator): one year treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sunitinib — one-year adjuvant Treatment with Sunitinib, schematic (4:2): 4 weeks (28) 50 mg(milligram) daily, 2 weeks (14) break
  Other Names: adjuvant Treatment
  Arms: Sunitinib
Drug: Placebo — one-year Treatment, schematic (4:2): 4 weeks (28) 50 mg(milligram) daily, 2 weeks (14) break,
  Other Names: Plazebo
  Arms: Placebo

SUMMARY:
The aim ist to identify biomarkers in the blood, to indicate early response or early treatment resistance.

DETAILED DESCRIPTION:
Prospective randomized multi-center Phase II trial for resection of metastases from pulmonary metastases (poor prognosis) in clear cell renal cell carcinoma + / - adjuvant sunitinib therapy over one year

ELIGIBILITY:
Inclusion Criteria:

* >/= 2 synchronous or within 24 Months after Nephrectomy occured pulmonary metastases. Patients in whom more back than 2 years of a solitary lung metastasis, bone metastasis or brain metastasis was resected, may also be included in the study.
* Aged 18 to 75 years
* functionally acceptable surgical risk
* Women in conceptional age: negative pregnancy test and adequate contraception
* Adequate hematologic, renal, hepatic and coagulation-physiological functions
* Amylase/ Lipase < 1,5 x upper limit of normal
* Informing the patient about the study and the present written consent to participate after clarification in accordance with the stipulations of AMG(german drug law), and the principles of GCP ("informed consent")
* Patient compliance and geographic proximity to allow adequate follow-up

Exclusion Criteria:

* Presence of other metastases outside the lung
* progress in the 12-week sunitinib therapy before resection of metastases
* R1 or R2-finding in resection of metastases
* Dialysis after nephrectomy
* Previous or existing serious cardiovascular (grade III - IV according to NYHA(New York Heart Association)) disease, active angina pectoris or ischemia, myocardial infarction within previous 6 months , uncontrolled hypertension(RR diastolic 120 mmHg(Millimeters of mercury))
* serious hematopoetic (e.g. serious Bone marrow aplasia), pulmonary, hepatic or renal Disease
* Stroke within the previous six months
* Patients with poorly controlled diabetes mellitus
* Serious bacterial or fungal infections
* chronic hepatitis B or C, HIV(human immunodeficiency virus) infection
* autoimmune disease
* prior organ transplantation
* prior autologous bone marrow transplant or stem cell transferred within the last 4 months before study
* Neuropsychiatric diseases that affect patient compliance
* Manifesto, second malignancy or other malignancy within the past 5 years (except basal cell carcinoma, carcinoma in situ of the cervix, incidental prostate carcinoma, superficial urothelial Ca pTaG1-2 and pT1G1)
* Therapy with immunotherapeutic agents including monoclonal antibodies, cytotoxic drugs or hormones (other than bisphosphonates and oral contraceptives) within the last 4 weeks prior to enrollment. Previous use of inhibitors of Ras/Raf-, MEK kinase, AKT kinase and mTOR inhibitors or induction of Farnesyltransferase
* Previous use of angiogenesis inhibitors such as VEGF / VEGFR, PDGF / PDGFR and other key molecules of angiogenesis
* parallel treatment with rifampicin
* Participation in other treatment studies in the last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
2 year relapse-free survival | 5 years

SECONDARY OUTCOMES:
perioperative mortality and morbidity | 5 years
Side effect of adjuvant therapy | 5 years
Quality of Life of the Patient | 5 years
Overall Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Krege, Priv. Doz. Dr. med., Principal Investigator — urological hospital of Maria Hilf Krankenhaus Krefeld
Locations (11):
- Germany (11):
  - Universitätsmedizin Charité Berlin, Berlin
  - Franziskus Krankenhaus, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - university hospital of Düsseldorf, Düsseldorf
  - university hospital of Essen, Essen
  - Ruhrlandklinik Department of Thoracic Surgery, Essen
  - university hospital of Freiburg, Freiburg im Breisgau
  - university Hospital of Heidelberg, Heidelberg
  - urological hospital of Maria Hilf Krankenhaus Krefeld, Krefeld
  - Hospital of Großhadern, München
  - Dr.-Horst-Schmidt-Kliniken GmbH, Wiesbaden